CLINICAL TRIAL: NCT00026013
Title: Effects of Hypericum Perforatum on Effectiveness of Oral Contraceptives
Brief Title: Effects of St. John's Wort on the Effectiveness of Oral Contraceptives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT000836-01 (NIH)
Record Dates: First submitted 2001-11-05; First posted 2001-11-06 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Contraception
Keywords: contraception; hormonal contraception; herbal remedies; hypericum perforatum; contraceptive effectiveness
MeSH Terms: interventions — Hypericum extract LI 160

INTERVENTIONS:
Drug: hypericum perforatum

SUMMARY:
The purpose of this study is to evaluate the effects of a common herbal remedy, St. John's Wort, on the effectiveness of birth control pills. St. John's Wort has recently been shown to increase metabolism of some drugs. If it could increase metabolism of oral contraceptives as well, it may increase the risk of contraceptive failure and unintended pregnancy. Study participants will be evaluated for risk of ovulation on oral contraceptives before and during simultaneous therapy with St. John's Wort.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Women taking or willing to take low dose oral contraceptives for 5 months
* No contraindications to hormonal contraception

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25
Dates: Start 2002-01; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Murphy, DrPh, Principal Investigator — Columbia University
Locations (1):
- Columbia University Department of Obstetrics & Gynecology, New York, New York, United States